CLINICAL TRIAL: NCT03671525
Title: Cognitive Effects of Nimodipine in Patients With Schizophrenia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00168634
Record Dates: First submitted 2018-08-06; First posted 2018-09-14 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia; Schizo Affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Nimodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nimodipine (Experimental): One 60mg capsule of nimodipine on first or second study visit
  Interventions: Drug: Nimodipine
- Placebo (Placebo Comparator): One placebo capsule on first or second study visit
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Nimodipine — Subject will receive two 30mg capsules of nimodipine during study visit.
  Other Names: Nymalize
  Arms: Nimodipine
Drug: Placebo oral capsule — Two coconut oil capsules that mimic the size and color of the nimodipine capsules
  Arms: Placebo

SUMMARY:
This study aims to evaluate the acute effects of nimodipine on cognitive performance in patients with schizophrenia using a battery of cognitive assessments.The subjects will also complete a 30-minute structural and functional MRI scan, with the goal of linking brain activity with working memory performance. Investigators predict that the performance increase induced by nimodipine will be greater in subjects who carry the A allele for the Calcium Voltage-Gated Channel Subunit Alpha1 C (CACNA1C) risk single nucleotide polymorphism (SNP) (rs1006737) in comparison to the response of G carriers.

DETAILED DESCRIPTION:
The main cognitive task of interest in this study is the N-back task because of the observed attenuation of prefrontal and parietal cortical activity after nimodipine administration in healthy subjects. Investigators hypothesize that acute nimodipine administration will improve cortical activation, which will lead to improved cognitive performance. The current study will provide insight whether nimodipine or another calcium channel blocker could be used as a treatment approach to alleviate cognitive deficits in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* This study will recruit patients with schizophrenia and/or schizoaffective disorder

Exclusion Criteria:

* past or current neurological disorder (including stroke, brain tumor, epilepsy, Alzheimer's, Parkinson's or Huntington's disease)
* uncontrolled medical disorder
* current or past hypotension
* head trauma with loss of consciousness in the last year or any evidence of functional impairment due to and persisting after head trauma
* positive pregnancy test, or currently breast feeding
* having an adverse reaction to nimodipine, or other calcium channel blocker

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Brain activity as assessed by BOLD fMRI | between 30 min and 1 hour after dose
  participants will complete an MRI scan to link brain activity with cognitive performance. Measures will be recorded in Arbitrary units.
Changes in Visual Learning and Memory Score | approximately an hour after dose
  Participants will complete the Brief Visuospatial Memory Task - Revised (BVMT-R) before and after administration of drug or placebo to determine the effect of nimodipine on visuospatial memory in patients with schizophrenia. Scores range from 0 to 60, with higher values indicating better performance. Administration takes approximately 45 minutes to complete (including a 25 minute delay)
Changes in Auditory Learning and Memory Score | approximately an hour after dose
  During each study visit, participants will complete the Hopkins Verbal Learning Task - Revised (HVLT-R) before and after administration of drug or placebo to determine the effect of nimodipine on verbal learning and memory in patients with schizophrenia. Scores range from 0 to 60, with higher values indicating better performance. Administration takes approximately 35 minutes to complete (including a 20-25 minute delay).
Changes in Global Neurocognitive effect as assessed by the Global Neurocognitive Assessment (GNA) | approximately an hour after dose
  During each study visit, participants will complete the Global Neurocognitive Assessment (GNA) before and after administration of drug or placebo to determine the effect of nimodipine on a range of neurocognitive measures in patients with schizophrenia. The GNA contains 10 items with varying score ranges. Higher scores indicate better performance.

SECONDARY OUTCOMES:
Effect of CACNA1C genotype on cognitive performance measures | during 2-3 hour study visit
  The CACNA1C risk-associated SNP (rs1006737) will be tested using a linear regression (with copy of A alleles) with each cognitive domain score to determine if CACNA1C genetics impact response to nimodipine.
Broader genetic associations with cognitive performance | during 2-3 hour study visit
  Genetic data will be used more broadly to include testing of the effects of genetic variation including but not limited to schizophrenia, cognition, behavior, and drug metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bigos, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland